CLINICAL TRIAL: NCT04204187
Title: Developing and Validating the Caring Questionnaire of Service Learning Courses: Using the Transformative Learning Model and Theory of Planned Behavior
Brief Title: Developing and Validating the Caring Questionnaire of Service Learning Courses
Status: Completed | Type: Observational
Sponsor: Central Taiwan University of Science and Technology (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Chiu Shu-Ching, assistant professor of nursing department, Central Taiwan University of Science and Technology
Other Study IDs: MOST 108-2637-B-166-002
Record Dates: First submitted 2019-12-15; First posted 2019-12-18 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: CARING; SERVICE LEARNING

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: service learning — service learning for university students

SUMMARY:
Research purposes: 1. Construct the caring scale in service learning courses. 2. Verify the reliability and validity of caring scale in service learning curriculum.

DETAILED DESCRIPTION:
Background: The core value of healthcare education is caring. However, caring traits are learned and acquired. Service learning advocates learning by doing. Through experience learning, students are guided to learn caring attitude or caring behaviour. Thus, teachers should construct appropriate assessments to understand caring traits as a transformative process from students' learning. Teachers should also adjust the pace of teaching continuously and design appropriate courses to facilitate students' achievement of their learning goals.

ELIGIBILITY:
Inclusion Criteria:

* undergraduate students after attending a service learning course

Exclusion Criteria:

* undergraduate students who refuse or are unwilling to participate in service learning courses.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: undergraduate students
Sampling Method: Probability Sample
Enrollment: 483 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2022-12-02 (Actual); Study Completion 2023-07-21 (Actual)

PRIMARY OUTCOMES:
first impression scale of service facility | up to 48 month
  Developing and validating the first impression scale in traditional Chinese language. The study uses the likert scale with five point scale: very positive, positive, neutral, negative, and very negative. The more positive feeling is more higher score.
service-learning experience of scale for caring | up to 48 month
  Developing and validating the service-learning experience scale for caring in traditional Chinese language. A higher score indicates more caring experiences.
organizational climate for service-learning | up to 48 month
  Developing and validating the organizational climate survey for service-learning in traditional Chinese language. The study uses the likert scale with five point scale: very positive, positive, neutral, negative, and very negative. The more positive feeling is more higher score.
idea transformation questionnaire for service-learning | up to 48 month
  Developing and validating a idea transformation questionnaire after service-learning in traditional Chinese language. A higher score indicates more idea changes.
perceived behavioral control for caring | up to 48 month
  Developing and validating the perceived behavioral control for caring in traditional Chinese language. The study uses the likert scale with five point scale: agree strongly, agree, neutral, disagree, and disagree strongly. The higher score indicates higher caring ability. The lower score indicates more difficult/limited to do caring behavior.
behavioral intention of caring | up to 48 month
  Developing and validating the behavioral intention of caring in traditional Chinese language. The study uses the likert scale with five point scale: agree strongly, agree, neutral, disagree, and disagree strongly. The higher score indicates higher commit for caring behavior in the near future.

SECONDARY OUTCOMES:
attitude of caring | after service-learning activity 1 month
  Three items for personal attitude towards caring including cognition, affection and behavior. The score range from 0-15. The higher score means more positive attitude of caring.
subjective norms | after service-learning activity 1 month
  Personal caring ability is mainly influenced by those important people. The study uses the likert scale with five point scale: very important, important, neutral, unimportant, and very unimportant. The more important feeling is more higher score.
selfishness questionnaire | after service-learning activity 1 month
  Validating and reliability for selfishness scale in traditional Chinese language. The range score is from 0-48. A higher score indicates more selfishness.

CONTACTS AND LOCATIONS:
Locations (1):
- Central Taiwan University of Science and Technology, Taichung, Taiwan